CLINICAL TRIAL: NCT05065918
Title: Text Message Intervention for Alcohol Use and Sexual Violence in College Students (STUDY00010873)
Brief Title: Text Message Intervention for Alcohol Use and Sexual Violence in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Pittsburgh (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 275726; K23AA027288 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-10-04 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use, Unspecified; Sexual Violence; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - alcohol use reduction content (Active Comparator): Alcohol use reduction content
  Interventions: Behavioral: alcohol use reduction content
- Intervention - sexual violence and alcohol use harm reduction content (Experimental): sexual violence and alcohol use harm reduction content
  Interventions: Behavioral: sexual violence and alcohol use harm reduction text message content

INTERVENTIONS:
Behavioral: sexual violence and alcohol use harm reduction text message content — The multi-target sexual violence harm reduction and alcohol use intervention will use a similar model to the alcohol use reduction intervention previous developed and implemented. Students will be: 1) queried via TM prior to typical drinking days regarding both alcohol use and SV harm reduction goal setting; 2) provided with goal reminders during drinking period; and 3) assessed for goal attainment and given feedback following drinking episodes. As with the control condition, post-drinking assessment happens weekly on Sundays. Monday thru Saturday participants will randomly receive or not receive one appropriate message pathway from the message library using the pre-determined pathways for messages.
  Arms: Intervention - sexual violence and alcohol use harm reduction content
Behavioral: alcohol use reduction content — The control condition will be a previously tested TM-delivered alcohol use reduction intervention. Prior to typical drinking occasions, individuals planning a drinking event are prompted to consider committing to a drinking limit goal, i.e.: "Would you be willing to set a goal to drink less than X drinks when drinking?". Based on willingness to commit to the goal, a feedback message is provided. During typical drinking periods, individuals receive a goal reminder. Each week, the program provides goal success/failure feedback or drinking quantity feedback. For example, those occasions where an individual committed to a drinking limit goal triggers either messages to reinforce goal successes or reframe goal failures. When an individual did not commit to a drink limit goal, they are provided feedback based on alcohol quantity (e.g. high risk drinking feedback).
  Arms: Control - alcohol use reduction content

SUMMARY:
This study is designed to pilot a text message (TM) delivered behavior change intervention to decrease binge drinking and to increase use of sexual violence (SV) harm reduction strategies among college students.

DETAILED DESCRIPTION:
This is a prospective, open-label, feasibility trial of a text message-delivered intervention designed to increase use of sexual violence harm reduction strategies and decrease alcohol use among college students.

In this research study, participants will:

* be asked to complete three surveys, one survey at the start of the study, one at the end of 3 month intervention period, and one at 6 months after enrollment
* receive one of two sets of text messages for a 3 month intervention period and be asked to respond to some of those text messages

  * Control condition text messages: The control condition will be a version of the TM-delivered alcohol use reduction intervention developed and implemented by Dr. Brian Suffoletto while at the University of Pittsburgh. This intervention has been tested in young adults (age 18-25) recruited from Emergency Department and college settings, and will be used to provide an attention control group for efficacy testing. Prior to typical drinking occasions, individuals planning a drinking event are prompted to consider committing to a drinking limit goal, i.e.: "Would you be willing to set a goal to drink less than X drinks when drinking?". Based on willingness to commit to the goal, a feedback message is provided. During typical drinking periods, individuals receive a goal reminder. Each week, the program provides goal success/failure feedback or drinking quantity feedback. For example, those occasions where an individual committed to a drinking limit goal triggers either messages to reinforce goal successes or reframe goal failures. When an individual did not commit to a drink limit goal, they are provided feedback based on alcohol quantity (e.g. abstinence feedback, high risk drinking feedback).
  * Intervention condition text messages: The multi-target sexual violence harm reduction and alcohol use intervention will use a similar model to the alcohol use reduction intervention previous developed and implemented at the University of Pittsburgh.13-15 Students will be: 1) queried via TM prior to typical drinking days regarding both alcohol use and SV harm reduction goal setting; 2) provided with goal reminders during drinking period; and 3) assessed for goal attainment and given feedback following drinking episodes.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-24 years,
2. current college or university student,
3. owns a mobile phone with internet access and unlimited text message plan,
4. reports binge drinking in the past 30 days [>3 drinks for women, >4 drinks men in one sitting]
5. Able to complete participation in English.
6. To evaluate messages tailored to prior SV victimization, approximately 50% of the sample will also be purposively recruited for a baseline history of SV.

Exclusion Criteria:

1. Under 18 years old, over 24 years old
2. Not currently enrolled in college
3. Does not own a mobile phone with internet access and unlimited data plan
4. Does not report binge drinking in the past 30 day
5. Unable to complete study participation in English

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Anderson, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Started | 92 | 91
Completed | 91 | 89
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 91 | 183
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (1.07) | 21 (1.47) | 20 (1.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 69 | 142
  Male | 19 | 22 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 87 | 83 | 170
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 73 | 73 | 146
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 92 | 91 | 183

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days Per Month
Description: as measured using a 30-day timeline follow-back (TLFB)
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: drinking days in the past 30 days
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 92 | 91
drinking days in the past 30 days | 6.45 (4.50) | 5.91 (4.97)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; Pilot sample size considerations: Assessing 70 students per arm (total n=140) that have completed the program and follow up would provide sufficient data on the full RCT protocol across multiple campuses as well as estimates of intervention effects. Assuming a retention rate of 70% for the three-month follow up, we would need to enroll 200 participants at baseline. We do not anticipate sufficient power to detect statistically and clinically significant results; Test type: Superiority; p = 0.448, Regression, Linear; Slope = -0.536, 95% CI 2-sided [-1.929 to 0.857]

2. Primary Outcome: Number of Drinking Days Per Month
Description: as measured using a 30-day timeline follow-back (TLFB)
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: drinking days in the past 30 days
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 91 | 89
drinking days in the past 30 days | 5.98 (3.84) | 6.00 (3.85)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.969, Regression, Linear; Slope = 0.99, 95% CI 2-sided [-1.152 to 1.108]

3. Primary Outcome: Number of Binge Drinking Days Per Month
Description: as measured using a 30-day timeline follow-back (TLFB)
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: binge drinking days in the past 30 days
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 92 | 91
binge drinking days in the past 30 days | 6.45 (4.50) | 5.91 (4.97)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.231, Regression, Linear; Slope = -0.5, 95% CI 2-sided [-1.322 to .322]

4. Primary Outcome: Number of Binge Drinking Days Per Month
Description: as measured using a 30-day timeline follow-back (TLFB)
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: binge drinking days in the past 30 days
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 91 | 89
binge drinking days in the past 30 days | 2.03 (2.55) | 1.71 (2.51)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.398, Regression, Linear; Slope = -0.319, 95% CI 2-sided [-1.064 to .425]

5. Primary Outcome: Use of Sexual Violence Harm Reduction Strategies
Description: Use of sexual violence harm reduction strategies assessed with an 11 item scale used by the American College Health Association's National College Health Survey of Protective Behavioral Strategies. Participants report on how often when drinking/socializing in the past 3 months they used each of the specific behaviors on a 5-point Likert scale ranging from (1 = never, 5 = always; theoretical range 11-55) with higher scores indicating higher frequency use of harm reduction strategies.
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 92 | 91
score on a scale | 36.72 (6.38) | 37.26 (6.19)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.382, Regression, Linear; Slope = 0.284, 95% CI 2-sided [-.356 to .924]

6. Primary Outcome: Use of Sexual Violence Harm Reduction Strategies
Description: as for outcome 5
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 91 | 89
score on a scale | 37.26 (6.19) | 36.20 (6.33)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.266, Regression, Linear; Slope = 0.382, 95% CI 2-sided [-.284 to 1.025]

7. Secondary Outcome: Knowledge of Sexual Violence and Alcohol Risk
Description: Alcohol and sexual consent scale. A series of questions were asked to measure recognition of what constitutes sexual violence and attitudes related to the role of alcohol in risk for sexual violence.
  12 item scale, using a 5-point Likert scale ranging from ("strongly disagree" to "strongly agree"; theoretical range of 12-60), with a higher mean score indicating greater knowledge and recognition.
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 92 | 91
score on a scale | 37.35 (3.95) | 36.72 (3.72)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; Test type: Superiority; p = 0.019, Regression, Linear; Slope = 0.530, 95% CI 2-sided [0.089 to .970]

8. Secondary Outcome: Knowledge of Sexual Violence and Alcohol Risk
Description: as for outcome 7
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 91 | 89
score on a scale | 37.11 (3.58) | 36.70 (5.51)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.284, Regression, Linear; Slope = 0.277, 95% CI 2-sided [-.232 to 0.787]

9. Secondary Outcome: Self-efficacy to Obtain Sexual Consent.
Description: Perceived behavioral control subscale of the Sexual Consent Scale-Revised. Participants reported how efficacious they feel at obtaining consent for sexual activity of a 5-point Likert scale. 11 item scale ("strongly disagree" to "strongly agree"; theoretical range of 11-55). Higher scores indicate greater self-efficacy.
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 92 | 91
score on a scale | 42.78 (7.03) | 40.92 (7.74)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.076, Regression, Linear; Slope = 0.709, 95% CI 2-sided [-.076 to 1.494]

10. Secondary Outcome: Self-efficacy to Obtain Sexual Consent.
Description: as for outcome 9
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
Number analyzed (Participants) | 91 | 88
score on a scale | 42.42 (7.29) | 40.53 (7.42)
Statistical Analysis 1: Comparison: Control - Alcohol Use Reduction Content vs Intervention - Sexual Violence and Alcohol Use Harm Reduction Content; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.136, Regression, Linear; Slope = 0.625, 95% CI 2-sided [-.199 to 1.449]

ADVERSE EVENTS:
Time Frame: Participants were followed for six months after enrollment/baseline data collection.
Arm/Group | Control - Alcohol Use Reduction Content | Intervention - Sexual Violence and Alcohol Use Harm Reduction Content
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 0/92 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT05065918/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT05065918/SAP_001.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05065918/ICF_002.pdf